CLINICAL TRIAL: NCT04221958
Title: Surface ECG Mapping in Healthy Adult Volunteers
Brief Title: Surface ECG Mapping
Status: Withdrawn | Type: Observational
Why Stopped: Unable to start the study due to changes in personnel.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Other Study IDs: 54619
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Electrocardiogram
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Electrocardiogram (ECG) Mapping: Participants will have 10 superficial electrode-patches placed on their chest in two vertical columns of 5 electrode-patches. The channels V1-V5 will be connected to one of the columns. The channel V6 will be connected to each of the electrode-patches in the second column ad recordings will be taken for approximately 2 minutes on each electrode-patch. ECG readings will be recorded.
  Interventions: Device: Electrocardiogram

INTERVENTIONS:
Device: Electrocardiogram — An electrocardiogram measures the electrical activity of the heartbeat. This "intervention" will be used on healthy adult volunteers whom are part of the staff at the institution.

SUMMARY:
This study aims to confirm a scientific concept that superficially placed electrocardiogram (ECG) leads may be compared to one another to help determine positioning. If proven to be effective, this could offer a more non-invasive means of positioning using superficial ECG tracings.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers from institution's staff
* Age >18 years

Exclusion Criteria:

- Existing heart conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of participants include healthy volunteers from the research/administrative/health care staff from the institution.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ECG Tracing | Approximately 30 minutes
  ECG tracing for each electrode will be recorded in voltage per unit of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States